CLINICAL TRIAL: NCT04283539
Title: Identification of Pathways to Mitigate Immune-Related Adverse Events With Cancer Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Jeffrey Kern, Professor of Medicine, National Jewish Health
Other Study IDs: ircAE HS-3411
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: checkpoint inhibitor; immuno-oncology; cutaneous adverse events
MeSH Terms: conditions — Neoplasms | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPI with ircAE: Participants on check point inhibitors with immune related cutaneous adverse event
  Interventions: Drug: systemic corticosteroid or biologic
- no ircAE: Participants who do not have a cutaneous adverse event

INTERVENTIONS:
Drug: systemic corticosteroid or biologic — Treatment with systemic corticosteroids or biologic therapies (for corticosteroid refractory patients or these in which corticosteroids are not the treatment of choice)
  Groups: CPI with ircAE

SUMMARY:
This protocol is a prospective, observational study of participants receiving immunotherapy (checkpoint inhibitors, CPI) for cancer therapy, testing the hypothesis that patients with immune related cutaneous adverse events (ircAEs) have unique immunologic endotypes associated with polarized immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, >18 yo
4. Diagnosis of solid tumor including, but not limited to, genitourinary/gynecologic, lung, gastrointestinal and melanoma
5. Receiving, or prior to starting on, a checkpoint inhibitor
6. Grade ≥ 2 ircAE (CTCAE v 5.0) (for cohort 1 only)
7. An indication for system corticosteroids or biologic therapies as determined by the treating physician (for cohort 1 only)
8. Life expectancy ≥ 12 weeks

Exclusion Criteria:

1. Daily use of systemic steroid treatment in the past 4 weeks (prednisone >10mg a day or equivalent) except for indications other than the cutaneous adverse event, and/or as an anti-emetic pre- or post-chemotherapy infusions.
2. Enrollment in any investigational drug trial with a drug that has not been approved
3. Taking other checkpoint inhibitors beyond anti-PD-(L)-1 or anti-CTLA-4 not yet indicated/approved for use
4. Pregnancy
5. Known blood borne infectious disease
6. Current or pervious diagnosis of a leukemia or lymphoma
7. Unable to give consent for study participation
8. Life expectancy < 12 weeks
9. Any other condition or diagnosis in the opinion of the investigator that would interfere with the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female with diagnosis of solid tumor
Sampling Method: Non-Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Immune Biomarkers | 30 days
  cytokines and chemokines

SECONDARY OUTCOMES:
Presence of skin and circulating lipid biomarkers which occur during and after ircAEs | 30 days
  Proportion of long-chain and short-chain ceramides Amounts and relative proportion of lysophosphatidylcholine molecular species. sphingosine-1-phosphate, platelet activating factor, leukotriene E4, prostaglandin F2α, endocannabinoids anandamide and 2- arachidonoylglycerol.
  Peripheral blood mononuclear cell RNA for expression of GRalpha, GRbeta, Vitamin D 24- Hydroxylase FK506 binding protein 5, mitogen induced kinase phosphatase 1, interleukin, tumor necrosis factor alphal
Mechanisms associated with corticosteroid unresponsiveness in patients with ircAE | 12 months
  Proportion of long-chain and short-chain ceramides Amounts and relative proportion of lysophosphatidylcholine molecular species. sphingosine-1-phosphate, platelet activating factor, leukotriene E4, prostaglandin F2α, endocannabinoids anandamide and 2- arachidonoylglycerol.
  Peripheral blood mononuclear cell RNA for expression of GRalpha, GRbeta, Vitamin D 24- Hydroxylase FK506 binding protein 5, mitogen induced kinase phosphatase 1, interleukin, tumor necrosis factor alphal

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - The Melanoma and Skin Cancer Institute, Denver, Colorado
  - Memorial Sloan Kettering Cancer Center, New York, New York